CLINICAL TRIAL: NCT04083924
Title: Preclinical Medical Student Handheld Echocardiography Training American Society of Echocardiography Curriculum
Brief Title: Preclinical Medical Student Echocardiography Training American Society of Echocardiography Curriculum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Responsible Party: Principal Investigator, Satoshi Jujo, Research Scholar, University of Hawaii
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-00265
Record Dates: First submitted 2019-09-03; First posted 2019-09-10 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Echocardiography; Medical Student; Transthoracic Echocardiography; Education
Keywords: Preclinical medical students; Handheld ultrasound; Butterfly iQ; Basic cardiac ultrasound; Focused cardiac ultrasound; Point of care; Training; Education; Flipped classroom

STUDY DESIGN:
Intervention Model Description: Pre-post education intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Basic cardiac ultrasound training (Experimental): Single group education intervention study. No control group. Pre-post educational outcomes only.
  Interventions: Other: Basic cardiac ultrasound training with Butterfly iQ handheld ultrasound

INTERVENTIONS:
Other: Basic cardiac ultrasound training with Butterfly iQ handheld ultrasound — Pre-training online module of the American society of Echocardiography and hands-on training of basic cardiac ultrasound with Butterfly iQ handheld ultrasound.

SUMMARY:
The investigators would like to evaluate how well pre-clinical medical students are able to perform a basic transthoracic echocardiography examination on a healthy volunteer using a hand-held ultrasound (HHU) after completing a flipped classroom echocardiography training methods which consist of pre-training e-learning, hands-on training, and competency assessment after the hands-on training.

DETAILED DESCRIPTION:
Background There is expanding need for cardiac ultrasound training for medical students, although most of medical schools do not integrate cardiac ultrasound training into their curricula. Most of residency programs already have some standardized cardiac ultrasound training for residents, but there is no standardized cardiac ultrasound training for medical students. Last year, the American Society of Echocardiography (ASE), which takes a leading role in establishing training for echocardiography, presented the recommended training methods of cardiac ultrasound for medical students with flipped classroom methods which consist of pre-training e-learning, hands-on training, and competency assessment after the hands-on training. But no researchers evaluated the effectiveness of the ASE recommended training methods at this moment. In addition, hand-held ultrasound (HHU) probe which enable us to perform echocardiography just connecting to cell phone, have become commercially available this year. The investigators believe most medical students will have their own HHU probe as well as physicians in ten years. Thus, the purpose of this study is to evaluate the ASE cardiac ultrasound training methods with applying the training methods to the pre-clinical medical students in University of Hawaii at Manoa using HHU probe.

Methods The investigators will perform a prospective, experimental educational study investigating the learning effects of ASE recommended echocardiography training in pre-clinical medical students on cognitive and psychomotor skill using HHU device, when performing a basic echocardiography on a healthy volunteer.

The investigators will use e-mail, presentations and public posting on bulletin board in University of Hawaii for recruiting participants of 1st or 2nd year medical students. Target sample size is 130 at maximum. After recruitment of participants, first, participants will take a pre-training knowledge assessment and questionnaire on basic cardiac ultrasound (30 minutes) one week before the day of hands-on training. Second, after the pre-training assessment, participants will independently review the 40 minute American Society of Echocardiography (ASE) recommended e-learning module (https://aseuniversity.org/ase/lessons/47) on basic cardiac ultrasound prior to the hands-on training day. Third, on the day of hands-on training, participants will take a pre-training skill assessment and receive hands-on training for basic cardiac ultrasound with a healthy volunteer (HV) (60 minutes). Immediately after the hands-on training, participants will complete a post-training knowledge and skill assessment on basic cardiac ultrasound with a HV and questionnaire about participants' experience (30 minutes). Finally participants will take another post-training knowledge & skill assessment on basic cardiac ultrasound and questionnaire about participants' experience eight weeks after the hands-on training day to assess retention of their knowledge and skills on basic cardiac ultrasound with a HV (30 minutes).

In this study, investigators plan to use HHU probe, named Butterfly iQ hand-held ultrasound, Butterfly Network, Inc.

The knowledge assessment contains 40 MCQs on 5 basic views. In the skill assessment, participants will be asked to obtain 5 basic views on a HV in 2 minutes per view and the images are to be video-recorded. After de-identification of obtained images, the image quality of 5 basic views will be assessed by three independent blinded assessors using image quality scoring system investigators devised. One of investigators will take a role of a HV for echocardiography throughout this study consistently.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be preclinical medical students (1st year or 2nd year) at John A. Burns School of Medicine, University of Hawaii.
* Participants are eligible after completion of 1st year medical student core cardiology curriculum at John A. Burns School of Medicine, University of Hawaii.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Image quality score change from pre-training to eight weeks after training. | Eight weeks after hands-on training.
  Image quality score of five basic cardiac ultrasound views assessed by predefined test scoring system. In the scoring system, each view is assessed excellent (2 points), acceptable (1 points), or poor (0 point) for clinical use. Summed, total score, thus, ranges from 0 to 10 points.

SECONDARY OUTCOMES:
Image quality score change from pre-training to immediately after training. | Immediately after hands-on training.
  Image quality score of five basic cardiac ultrasound views assessed by predefined test scoring system. In the scoring system, each view is assessed excellent (2 points), acceptable (1 points), or poor (0 point) for clinical use. Summed, total score, thus, ranges from 0 to 10 points.
Knowledge test score change from pre-training to eight weeks after training. | Eight weeks after hands-on training.
  40 multiple choice questions about anatomical knowledge of five basic cardiac ultrasound views using Google Form. Total score ranges from 0 to 40 points.
Knowledge test score change from pre-training to immediately after training. | Immediately after hands-on training.
  40 multiple choice questions about anatomical knowledge of five basic cardiac ultrasound views using Google Form. Total score ranges from 0 to 40 points.
Overall 5-point Likert scale participants training satisfaction | Immediately after hands-on training.
  Overall participants training satisfaction assessed with 5-point Likert scale. This scale ranges from 1 to 5. Higher Likert scale represents higher participant training satisfaction.
Overall 5-point Likert scale participants training satisfaction | Eight weeks after hands-on training.
  Overall participants training satisfaction assessed with 5-point Likert scale. This scale ranges from 1 to 5. Higher Likert scale represents higher participant training satisfaction.
Participant confidence in basic cardiac ultrasound. | Immediately before hands-on training.
  Participant confidence in basic cardiac ultrasound assessed with 5-point Likert scale. This scale ranges from 1 to 5. Higher Likert scale represents higher participants confidence in basic cardiac ultrasound.
Participant confidence in basic cardiac ultrasound. | Immediately after hands-on training.
  Participant confidence in basic cardiac ultrasound assessed with 5-point Likert scale. This scale ranges from 1 to 5. Higher Likert scale represents higher participants confidence in basic cardiac ultrasound.
Participant confidence in basic cardiac ultrasound. | Eight weeks after hands-on training.
  Participant confidence in basic cardiac ultrasound assessed with 5-point Likert scale. This scale ranges from 1 to 5. Higher Likert scale represents higher participants confidence in basic cardiac ultrasound.
Findings of post-training predefined survey | Immediately after hands-on training.
  Findings of post-training predefined survey regarding usefulness of training.
Findings of post-training predefined survey | Eight weeks after hands-on training.
  Findings of post-training predefined survey regarding usefulness of training.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Berg, MD, Study Director — SimTiki Simulation Center, John A. Burns School of Medicine.
Locations (1):
- SimTiki Simulation Center, John A. Burns school of medicine, University of Hawaii at Manoa, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johri AM, Durbin J, Newbigging J, Tanzola R, Chow R, De S, Tam J. Cardiac Point-of-Care Ultrasound: State-of-the-Art in Medical School Education. J Am Soc Echocardiogr. 2018 Jul;31(7):749-760. doi: 10.1016/j.echo.2018.01.014. Epub 2018 Mar 15. PMID 29550326
- [Derived] Jujo S, Lee-Jayaram JJ, Sakka BI, Nakahira A, Kataoka A, Izumo M, Kusunose K, Athinartrattanapong N, Oikawa S, Berg BW. Pre-clinical medical student cardiac point-of-care ultrasound curriculum based on the American Society of Echocardiography recommendations: a pilot and feasibility study. Pilot Feasibility Stud. 2021 Sep 14;7(1):175. doi: 10.1186/s40814-021-00910-3. PMID 34521479
- See also: Online training module for Cardiovascular Point-of-Care Imaging for the Medical Student and Novice User on American Society of Echocardiography web site — https://aseuniversity.org/ase/lessons/47